CLINICAL TRIAL: NCT00926146
Title: HBV Prevention for Homeless at Risk for HBV/HCV/HIV
Brief Title: Hepatitis B Virus (HBV) Prevention for Homeless at Risk for HBV/Hepatitis C Virus (HCV)/HIV
Acronym: HBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, PhD, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 090602901; DA016147 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis B; Hepatitis C; HIV; HIV Infections
Keywords: Hepatitis B and C; HIV; nurse case management; HIV seronegativity
MeSH Terms: conditions — Hepatitis B; Hepatitis C; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCMIT (Experimental): Nurse Case Management Plus Contingency Management and Tracking and the HBV vaccine
  Interventions: Behavioral: NCMIT
- SCMIT (Active Comparator): Standard with Contingency Management and Tracking (SCMT) and HBV vaccine
  Interventions: Behavioral: SCMIT

INTERVENTIONS:
Behavioral: NCMIT — Nurse Case Management Plus Contingency Management and Tracking (NCCMT) Program includes 20 minute case management, delivered by the NCCMT nurse and a separate 45 minute culturally competent specialized education, delivered by the two assigned nurses and research assistants weekly over 8 weeks. Participants of this group will also receive the HBV vaccine subsequently at one month and four months after baseline and incentives for three-weekly urine samples.
  Arms: NCMIT
Behavioral: SCMIT — Standard with Contingency Management and Tracking (SCMT) Program. Participants in the SCMT group will interact three times a week over the four-month intervention period with the research nurse and research assistant and will be offered: 1) a brief HBV/HCV education program; 2) receipt of the vaccine subsequently at one month and four months after baseline; and 3) voucher incentives for three-weekly urine samples. The SCMT participants will not receive the specialized education sessions nor the case management delivered weekly over the first 8 weeks sessions.
  Arms: SCMIT

SUMMARY:
In this study, researchers from UCLA and Friends Community Center will work together in designing a program to assist young homeless stimulant-using gay and bisexual homeless men to complete the hepatitis vaccine and in reducing drug and sexual activity. Using nurse case management strategies, found successful with homeless adults as well as contingency management strategies, found successful with gay and bisexual homeless adults by the community partners, the investigators will evaluate the effectiveness of a program that combines both strategies. As stimulant use threatens to increase homeless persons' risk of exposure to hepatitis A and B viruses, particularly among young users who may not yet be HBV-infected, this research is targeted to engage this group in treatment, until they are suitably protected from HBV, and hopefully reduce risk for HCV and HIV as well.

DETAILED DESCRIPTION:
Homeless adults are at high risk for Hepatitis B virus (HBV), Hepatitis C virus (HCV) and HIV infection due to high rates of injection drug use and unprotected sexual activity. Our NIDA-funded RO1 award has enabled us to implement a successful intervention designed to evaluate the effectiveness of a HBV vaccination intervention with homeless adults. Our findings revealed that a greater percent of homeless adults randomized to the Nurse Case Managed Plus Incentive and Tracking group completed the HAV/HBV vaccine series compared to a Standard program without tracking. Homeless persons least likely to complete the vaccine series were young (< 40), and were men having sex with men (MSM); a significant number of these young adults also reported methamphetamine (MA) and cocaine/crack use. Stimulants (SAs), including MA and cocaine/crack are commonly used by homeless MSM, who contend with disorganized lives, unemployment, and little access to health and social services; thus, HBV vaccination is particularly challenging in this population. HAV/HBV vaccination and effective behavioral treatment are two of the most important strategies for reducing HBV infection among this at-risk group of SA users.

Based upon advice from our community partners who have successfully treated SA-using gay and bisexual men (GBM), we will incorporate contingency management into our vaccination completion program, which had lower completion rates among young adults and MSMs. Thus, in this competitive renewal, we propose a randomized, experimental, two-group design to evaluate the effectiveness of a Nurse Case Managed Program, which includes specialized education and Contingency Management and Tracking (NCCMT), with a Standard Program, including brief education, Contingency Management and Tracking (SCMT) with 500 homeless, young (18-39), SA-using GBM, on completion of the Twinrix HAV/HBV vaccine and, secondarily, on reduction of risk for hepatitis and HIV. This study is innovative in that it will allow us to look at the effect of an enhanced case management and contingency management program versus a standard contingency management program. The proposed study combines optimal strategies to approach, engage and intervene with a hidden and high-risk population to assess the feasibility and efficacy of interventions that may prove beneficial in preventing HBV and HAV infections. We will also assess the relative cost of these programs in terms of completion of the HAV/HBV vaccination series. As use of SAs threatens to intensify homeless persons' risk of exposure to HAV and HBV, particularly among young users who may not yet be HBV-infected, research targeted to engage this group in treatment, until they are suitably protected from HBV, is critical.

ELIGIBILITY:
Inclusion Criteria:

1. homeless males self-reporting gay or bisexual behaviors in the last 12 months
2. age 18-39
3. methamphetamine and/or cocaine/crack use currently or in the last three months
4. no self-reported participation in drug treatment in the last 30 days
5. willing to provide informed consent
6. willing to undergo hepatitis B and C and HIV antibody testing at baseline
7. found to be HBV antibody negative

Exclusion Criteria:

1. persons with Guillian Barre, or allergy to yeast or neomycin
2. monolingual speakers of languages other than English or Spanish
3. persons judged to be cognitively impaired by the nurse

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Compare the NCMIT and SCMT programs among homeless young gay and bisexual stimulant using men with respect to completion of a HBV vaccination series administered in three doses over a four-month period. | 5 years

SECONDARY OUTCOMES:
Document the occurrences of HCV and HIV infections as baseline among these homeless HBV antibody negative stimulant users, and the factors associated with these infections at baseline. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Nyamathi, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Friends Community Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyamathi A, Shoptaw S, Cohen A, Greengold B, Nyamathi K, Marfisee M, de Castro V, Khalilifard F, George D, Leake B. Effect of motivational interviewing on reduction of alcohol use. Drug Alcohol Depend. 2010 Feb 1;107(1):23-30. doi: 10.1016/j.drugalcdep.2009.08.021. PMID 19836904
- [Derived] Nyamathi A, Reback CJ, Shoptaw S, Salem BE, Zhang S, Yadav K. Impact of Tailored Interventions to Reduce Drug Use and Sexual Risk Behaviors Among Homeless Gay and Bisexual Men. Am J Mens Health. 2017 Mar;11(2):208-220. doi: 10.1177/1557988315590837. Epub 2016 Jul 8. PMID 26130725
- [Derived] Nyamathi AM, Nandy K, Greengold B, Marfisee M, Khalilifard F, Cohen A, Leake B. Effectiveness of intervention on improvement of drug use among methadone maintained adults. J Addict Dis. 2011 Jan;30(1):6-16. doi: 10.1080/10550887.2010.531669. PMID 21218306